CLINICAL TRIAL: NCT05695235
Title: Monitoring Sleep, Wellbeing, and Glucose Metabolism in Postgraduate Year 1 Doctors on Traditional and Float Call Shifts
Brief Title: Monitoring Sleep, Wellbeing, and Glucose Metabolism in PGY1s
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Michael W.L. Chee, Professor, National University of Singapore
Other Study IDs: NUHSsleepstudy
Record Dates: First submitted 2022-12-27; First posted 2023-01-23 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Sleep; Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traditional call: In the traditional overnight on-call system, each resident is on call for 4-6 nights per month (7 am - 5 pm, followed by overnight call until 8 am the next morning)
  Interventions: Device: CGM; Device: Oura ring; Behavioral: Cognitive tasks and questionnaires
- Float call: In the night float system, residents work from 8 pm to 8 am for 5 - 7 consecutive nights once every month
  Interventions: Device: CGM; Device: Oura ring; Behavioral: Cognitive tasks and questionnaires

INTERVENTIONS:
Device: CGM — Wearable continuous glucose monitoring systems (CGMS) provide a minimally invasive means of passively tracking ambulant interstitial fluid glucose levels in real time.
Device: Oura ring — Wearable sleep tracking device
Behavioral: Cognitive tasks and questionnaires — Participants will be prompted daily to fill out a short set of wellbeing questions and perform a short alertness test on their mobile phones and laptop.

SUMMARY:
Overnight on-call schedules can impact sleep, wellbeing, and alertness, which can be detrimental on the performance, physical and mental health of residents. Moreover, rotating shift work may have a long-term negative health impact (e.g. increased risk of diabetes). Within the National University Hospital (NUH), two different systems of rotating on-call schedules are implemented. In the night float system, residents work from 8 pm to 8 am for 5 - 7 consecutive nights once every month, compared to the traditional overnight on-call system, where each resident is on call for 4-6 nights per month (7 am - 5 pm, followed by overnight call until 8 am the next morning). The aim of the current study is to track sleep, wellbeing, and glucose metabolism during the different phases of the night float and traditional on-call schedules.

DETAILED DESCRIPTION:
Overnight on-call schedules can impact sleep, wellbeing, and alertness, which can be detrimental on the performance, physical and mental health of residents. Moreover, rotating shift work may have a long-term negative health impact (e.g. increased risk of diabetes). Within the National University Hospital (NUH), two different systems of rotating on-call schedules are implemented. In the night float system, residents work from 8 pm to 8 am for 5 - 7 consecutive nights once every month, compared to the traditional overnight on-call system, where each resident is on call for 4-6 nights per month (7 am - 5 pm, followed by overnight call until 8 am the next morning). The aim of the current study is to track sleep, wellbeing, and glucose metabolism during the different phases of the night float and traditional on-call schedules.

The availability of accurate mobile methodologies to monitor sleep and metabolic health provide new avenues for the improvement of sleep health and well-being. Wearable sleep tracking devices and smartphone apps provide remarkable opportunities for non-invasive, longitudinal sleep detection. Measurement of sleep during different stages of the shift schedule (baseline, on-call, recovery) can provide detailed insights into the temporal impact of the different schedules. Moreover, self-reported ratings of sleep quality, wellbeing, and time-use (delivered through phone-based e-diary methods) can further detail the mental health impact associated with these schedules.

Wearable continuous glucose monitoring systems (CGMS) provide a minimally invasive means of passively tracking ambulant interstitial fluid glucose levels in real time.

ELIGIBILITY:
Inclusion Criteria:

* NUHS Postgraduate year 1 doctors
* Above 21 years of age
* Completing their year 1 rotations in 2021 or 2022

Exclusion Criteria:

* As this is an observational study with minimal risk, in an restricted pool of participants, no further exclusion criteria will be applied for participation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NUHS Postgraduate year 1 doctors
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Sleep | 8 weeks
  Sleep duration and timing will be measured
Wellbeing | 8 weeks
  Participants will complete a daily micro questionnaire delivered through a mobile phone-based application. The investigators will examine mood ratings and stress ratings. Participants will be asked to respond to questions such as "How are you feeling right now?", rating their response from 'Negative' to 'Positive' on a 100-points sliding bar, "How stressed are you feeling right now?", rating their response from 'Not at all stressed' to 'Very stressed' on a 100-points sliding bar.
Glucose monitoring | 2 weeks
  Blood glucose will be recorded using a wearable continuous glucose monitoring sensor (CGM: FreeStyle Libre Pro iQ by Abbott). CGM period will be individually scheduled to coincide with at least one cycle of day shift-night shift- recovery for each participant.
Alertness | 8 weeks
  Participants will complete a daily set of cognitive games, delivered through a mobile phone-based application. The outcome measure from the games is a 3-min psychomotor vigilance task measuring sustained attention. Specifically, the investigators examine median reaction time and lapses (reaction time > 500ms).

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, (No States Listed), Singapore

IPD SHARING:
Plan to Share IPD: No